CLINICAL TRIAL: NCT04310059
Title: A Randomized Controlled Trial to Study the Effect of Folic Acid Supplementation in Pregnant Women Having Thalassaemia Trait
Brief Title: Effect of Folic Acid Supplementation in Pregnant Women Having Thalassaemia Trait
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Queen Mary Hospital, Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UW 20-084
Record Dates: First submitted 2020-03-05; First posted 2020-03-17 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Thalassemia; Folic Acid Deficiency Anemia
MeSH Terms: conditions — Thalassemia | interventions — Folic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Folic acid 5mg (Active Comparator)
  Interventions: Dietary Supplement: Folic acid
- Folic acid 0.5mg (Active Comparator)
  Interventions: Dietary Supplement: Folic acid
- Materna (Active Comparator)
  Interventions: Dietary Supplement: Materna

INTERVENTIONS:
Dietary Supplement: Folic acid — women will be randomised into one of the three groups. Group A - Folic acid 5mg/day Group B - Folic acid 0.5mg/day Group C - Materna one tablet/day (a pregnancy supplement containing 0.6mg folic acid)
  Arms: Folic acid 0.5mg; Folic acid 5mg
Dietary Supplement: Materna — Materna
  Arms: Materna

SUMMARY:
Folic acid supplementation has been recommended for prevention of neural tube defects in pregnancy when taken periconceptionally up to 12 weeks of gestation. A daily dose of 0.4mg has been endorsed by World Health Organisation to achieve a Red blood cell (RBC) folate level of 906nmol/L (400ng/mL) for reduction of neural tube defect. Hong Kong has no policy on food fortification. Research data conducted in countries with food fortification may not be applicable. It is therefore essential to study the baseline folate status in pregnant women locally.

For pregnant women with thalassaemia, they are believed to have a higher risk of folate deficiency because of an increased rate of erythropoiesis and chronic haemolysis. However, information on folate level of thalassaemia trait in pregnancy is scanty. Unmetabolized folic acid has been detected in maternal and fetal blood when daily dosage greater than 0.8-1mg was taken. In term of the dosage and duration of folic acid supplementation after 12 weeks of gestation, the practice varies widely among public hospitals and Maternity & Child Health Care centres. It is therefore essential to study the optimal dosage of folic acid supplementation in women with thalassaemia.

DETAILED DESCRIPTION:
Folic acid supplementation is well established for its role in prevention of neural tube defects (NTD) when taken periconceptionally up to 12 weeks of gestation. The naturally occurring form, folate, is a water soluble B vitamin (B9) that is mostly present in dark green leafy vegetables and legumes. However, it is only 50% bioavailable. Folic acid, on the contrary, as a synthetic form of folate is almost completely bioavailable especially when administered in an empty stomach. It has been endorsed by World Health Organisation that RBC folate cutoff of 906 nmol/L (400ng/mL) is required for reduction of NTD. This level is only achievable by taking Folic acid supplementation of 0.4mg/day. Women at higher risk of having recurrent NTD is recommended to take higher dose at 4mg/day.

Patients with thalassaemia have an increased rate of erythropoiesis and chronic haemolysis. They are believed to have a higher rate of folate turnover and consequentially higher risk of folate deficiency. Guideline from Royal College of Obstetricians and Gynaecologists recommends daily intake of 5mg folic acid preconceptionally to prevent NTD. But, it does not specify whether this dosage is applicable to all types and degrees of thalassaemias and research data on the optimal dosage is lacking.

In addition to prevention of NTD, the supplementation of folic acid is also recommended for pregnant thalassaemia women for prevention of antenatal anaemia. In a retrospective study of Chinese population reported in 1989, women with beta-thalassaemia minor taking additional 5mg folic acid had higher pre-delivery haemoglobin concentration of 10.1 g/dL compared to haemoglobin level of 9.7 g/dL in the group taking Obimin (a pregnancy supplement containing 0.25mg folic acid and 90 mg ferrous fumarate). However, there was no further randomised controlled trial to validate this observation. Though a higher folic acid supplementation was believed to be beneficial in prevention of antenatal anaemia, unmetabolized folic acid were detected in maternal and fetal blood when daily dosage greater than 0.8-1mg was taken. Moreover, a higher rate of urinary excretion of folic acid was also observed in pregnant women receiving higher dosage of folic acid supplementation.

In non-pregnant beta thalassaemia major patients, folic acid supplementation at 1 mg daily was advised as cessation of which could lead to a significant reduction in serum folate. This has been counter-proposed by the observation of normal to high serum folate levels in transfusion dependent thalassaemia receiving optimal transfusion. Indeed, folic acid supplementation should be considered for non-transfusion dependent thalassaemia as excessive erythropoiesis is required to maintain satisfactory haemoglobin.

Folate level drops during pregnancy to puerperal period. Information on folate level of thalassaemia trait in pregnancy is scanty. In a paper published in 1985, no difference in serum folate was found between normal women and women with thalassaemia trait, and hence usual supplementation was suggested.

Hong Kong has no policy on food fortification. Research data conducted in countries with food fortification may not be applicable. The folate status may have been changed in last few decades because of better general nutritional status and public knowledge of preconception folic acid supplementation. The preparation of 5mg folic acid is available in all public hospitals and preparation of 0.5mg folic acid is recently introduced. As such, the 5mg folic acid prescription is traditionally adopted and this can be a result of its availability. However, the practice varies widely among public hospitals and Maternity & Child Health Care centres. There is no standardised guideline on the dosage and indications of folic acid supplementation for pregnant thalassaemic women. More importantly, no recent data on the baseline folate status in pregnant women with thalassaemia is available locally.

Patient blood management in Obstetrics has been advocated with an aim to minimize blood loss by maintaining haemoglobin levels, reduce blood transfusion and optimize patient outcome. Identification and treatment of maternal anaemia is one of the three main pillars to achieve it. Even though thalassaemia can be considered as a risk factor for NTD, it remains controversial as to how much folic acid supplementation is adequate for pregnant women with thalassaemia trait in prevention of maternal anaemia which is a key element in maternity care.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy
* Alpha thalassaemia trait
* Beta thalassaemia trait

Exclusion Criteria:

* Women taking over 0.6mg folic acid daily for 3 months or more prior to and during pregnancy
* Gestational age > 16 weeks at first antenatal visit
* Women age =< 18 years old
* Booking BMI =< 18 or >= 35
* Serum ferritin level < 30ug/L or 68 pmol/L
* Concomitant alpha and beta thalassaemia
* Hb H disease
* Beta thalassaemia major
* Beta thalassaemia intermediate
* Thalassaemia other than alpha or beta type
* Women on long term medications
* Women with risk factors for NTD
* Women with known epilepsy
* Women with bariatric surgery or malabsorption diseases
* Women with known MTHFR polymorphism
* Vegetarian

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Only pregnant women are recruited
Enrollment: 270 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2025-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Haemoglobin level | Change in level throughout the pregnancy, up to 42 weeks
Maternal RBC folate concentration | Change in level throughout the pregnancy, up to 42 weeks
Maternal serum folate concentration | Change in level throughout the pregnancy, up to 42 weeks
Cord blood RBC | Upon birth
Cord blood serum folate concentration | Upon birth

SECONDARY OUTCOMES:
Ferritin level | Change in level throughout the pregnancy, up to 42 weeks
Maternal Vitamin B12 | Maternal Vitamin B12 at first antenatal visit
Cord blood vitamin B12 | Cord blood vitamin B12 upon birth

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Daly LE, Kirke PN, Molloy A, Weir DG, Scott JM. Folate levels and neural tube defects. Implications for prevention. JAMA. 1995 Dec 6;274(21):1698-702. doi: 10.1001/jama.1995.03530210052030. PMID 7474275
- [Background] Czeizel AE, Dudas I. Prevention of the first occurrence of neural-tube defects by periconceptional vitamin supplementation. N Engl J Med. 1992 Dec 24;327(26):1832-5. doi: 10.1056/NEJM199212243272602. PMID 1307234
- [Background] Crider KS, Devine O, Hao L, Dowling NF, Li S, Molloy AM, Li Z, Zhu J, Berry RJ. Population red blood cell folate concentrations for prevention of neural tube defects: Bayesian model. BMJ. 2014 Jul 29;349:g4554. doi: 10.1136/bmj.g4554. PMID 25073783
- [Background] US Preventive Services Task Force; Bibbins-Domingo K, Grossman DC, Curry SJ, Davidson KW, Epling JW Jr, Garcia FA, Kemper AR, Krist AH, Kurth AE, Landefeld CS, Mangione CM, Phillips WR, Phipps MG, Pignone MP, Silverstein M, Tseng CW. Folic Acid Supplementation for the Prevention of Neural Tube Defects: US Preventive Services Task Force Recommendation Statement. JAMA. 2017 Jan 10;317(2):183-189. doi: 10.1001/jama.2016.19438. PMID 28097362
- [Background] Cordero AM, Crider KS, Rogers LM, Cannon MJ, Berry RJ. Optimal serum and red blood cell folate concentrations in women of reproductive age for prevention of neural tube defects: World Health Organization guidelines. MMWR Morb Mortal Wkly Rep. 2015 Apr 24;64(15):421-3. PMID 25905896
- [Background] Prevention of neural tube defects: results of the Medical Research Council Vitamin Study. MRC Vitamin Study Research Group. Lancet. 1991 Jul 20;338(8760):131-7. PMID 1677062
- [Background] Management of Beta Thalassaemia in Pregnancy. Green-top Guideline No 66: Royal College of Obstetricians & Gynaecologists; 2014. p. 1-17.
- [Background] Lao TT. Obstetric care for women with thalassemia. Best Pract Res Clin Obstet Gynaecol. 2017 Feb;39:89-100. doi: 10.1016/j.bpobgyn.2016.09.002. Epub 2016 Sep 23. PMID 28341055
- [Background] Leung CF, Lao TT, Chang AM. Effect of folate supplement on pregnant women with beta-thalassaemia minor. Eur J Obstet Gynecol Reprod Biol. 1989 Dec;33(3):209-13. doi: 10.1016/0028-2243(89)90131-7. PMID 2599250
- [Background] Plumptre L, Masih SP, Ly A, Aufreiter S, Sohn KJ, Croxford R, Lausman AY, Berger H, O'Connor DL, Kim YI. High concentrations of folate and unmetabolized folic acid in a cohort of pregnant Canadian women and umbilical cord blood. Am J Clin Nutr. 2015 Oct;102(4):848-57. doi: 10.3945/ajcn.115.110783. Epub 2015 Aug 12. PMID 26269367
- [Background] Caudill MA, Cruz AC, Gregory JF 3rd, Hutson AD, Bailey LB. Folate status response to controlled folate intake in pregnant women. J Nutr. 1997 Dec;127(12):2363-70. doi: 10.1093/jn/127.12.2363. PMID 9405587
- [Background] Baghersalimi A, Hemmati Kolachahi H, Darbandi B, Kamran Mavardiani Z, Alizadeh Alinodehi M, Dalili S, Hassanzadeh Rad A. Assessment of Serum Folic Acid and Homocysteine in Thalassemia Major Patients Before and After Folic Acid Supplement Cessation. J Pediatr Hematol Oncol. 2018 Oct;40(7):504-507. doi: 10.1097/MPH.0000000000001295. PMID 30124548
- [Background] Tripathi G, Kalra M, Mahajan A. Folate supplementation in transfusion-dependent thalassemia: Do we really need such high doses? Indian J Med Paediatr Oncol. 2016 Oct-Dec;37(4):305. doi: 10.4103/0971-5851.195746. No abstract available. PMID 28144102
- [Background] Tso SC, Wong RL. Folate status in pregnant Chinese women in Hong Kong. Int J Gynaecol Obstet. 1980;18(4):290-4. doi: 10.1002/j.1879-3479.1980.tb00498.x. PMID 6109674
- [Background] White JM, Richards R, Byrne M, Buchanan T, White YS, Jelenski G. Thalassaemia trait and pregnancy. J Clin Pathol. 1985 Jul;38(7):810-7. doi: 10.1136/jcp.38.7.810. PMID 4019802
- [Background] Guideline: Fortification of Rice with Vitamins and Minerals as a Public Health Strategy. Geneva: World Health Organization; 2018. Available from http://www.ncbi.nlm.nih.gov/books/NBK531762/ PMID 30307723
- [Background] Atta CA, Fiest KM, Frolkis AD, Jette N, Pringsheim T, St Germaine-Smith C, Rajapakse T, Kaplan GG, Metcalfe A. Global Birth Prevalence of Spina Bifida by Folic Acid Fortification Status: A Systematic Review and Meta-Analysis. Am J Public Health. 2016 Jan;106(1):e24-34. doi: 10.2105/AJPH.2015.302902. Epub 2015 Nov 12. PMID 26562127
- [Background] Joseph CA, Dedman D, Fern K, Chakraverty P, Watson JM. Influenza surveillance in England and Wales: November 1991-June 1992. Commun Dis Rep CDR Rev. 1992 Dec 4;2(13):R149-52. No abstract available. PMID 1285133
- [Background] Gilchrest BA, Rowe JW, Brown RS, Steinman TI, Arndt KA. Relief of uremic pruritus with ultraviolet phototherapy. N Engl J Med. 1977 Jul 21;297(3):136-8. doi: 10.1056/NEJM197707212970304. PMID 865585